CLINICAL TRIAL: NCT01150344
Title: Effectiveness and Safety Evaluation of the Riamet® Versus Malarone® in the Treatment of Uncomplicated Malaria : a Multicentric Study
Brief Title: Evaluation of the Riamet® Versus Malarone® in the Treatment of Uncomplicated Malaria
Acronym: MalaRia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P081222; 2010-019950-42 (EudraCT Number)
Record Dates: First submitted 2010-06-18; First posted 2010-06-24 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-10

CONDITIONS: Malaria
Keywords: Multicentric study; Antimalarial; P. falciparum; Efficacy; Failures; Malarone; RIAMET
MeSH Terms: conditions — Malaria | interventions — atovaquone, proguanil drug combination; Atovaquone; Artemether

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Malarone (Active Comparator): Malarone (atovaquone + proguanil combination):
  patients treated with Malarone®
  Interventions: Drug: Malarone (atovaquone + proguanil combination)
- Riamet (Active Comparator): RIAMET (artemether + LUMEFANTRIN combination):
  patients treated with Riamet®
  Interventions: Drug: RIAMET (artemether + LUMEFANTRIN combination)

INTERVENTIONS:
Drug: Malarone (atovaquone + proguanil combination) — 4 X (250mg atovaquone + 100 mg proguanil) per os, once a day on 3 days as H0, H24 and H48.
  Other Names: atovaquone+proguanil combination
  Arms: Malarone
Drug: RIAMET (artemether + LUMEFANTRIN combination) — 4 X (20mg artemether + 120 mg lumefantrine) per os twice a day on 3 days as H0, H8, H24, H36, H48 and H60
  Other Names: artemether+LUMEFANTRIN combination
  Arms: Riamet

SUMMARY:
Riamet® or Malarone® are both recommended as the first line treatment for uncomplicated malaria in France, according to the French consensus Conference revised in 2007 on the treatment of imported malaria.

The aim of the study is to compare both tolerance and efficacy of Malarone® and Riamet® in the treatment of uncomplicated imported malaria and to determine clinical and parasitological predictive factors associated with a less effectiveness. It's a multicentric, randomised study in adults with uncomplicated malaria. Treatment will be administered for 3 days, and patients will be followed for 28 days, to evaluate the therapeutic evolution. 640 patients will be included among 15 centres.

DETAILED DESCRIPTION:
Background : RIAMET® or Malarone® are both recommended as the first line treatment for uncomplicated malaria in France, according to the French consensus Conference revised in 2007 on the treatment of imported malaria. Today no randomized controlled trial (RCT) comparing both treatments are available for either tolerance or efficacy especially in the field of imported malaria.

Malarone®, an atovaquone+proguanil combination, has become these last years the most prescribed treatment in adult in this indication in France. With Malarone®, therapeutic failures are rare, but digestive side effects are observed, such as vomiting, possibly leading to the use of a second line treatment.

Riamet®, an artemether+lumefantrine combination, is available in France since only July 2007, but is largely used in endemic areas (as CO-ARTEM). A good tolerance and efficacy are reported by studies performed in endemic areas.

Both antimalarials are to be taken for a 3-days treatment period, once a day for Malarone®, but twice a day for Riamet®, which is supposed to affect the observance, on the one hand. On the other hand, parasitological cure rate and apyrexia occur faster with RIAMETt® than with Malarone®.

Primary objective: to compare both tolerance et efficacy of Malarone® and RIAMET® in the treatment of uncomplicated imported malaria.

Secondary objective: to determine clinical and parasitological predictive factors associated with a less effectiveness.

Primary outcome: Number of cases where a second line treatment is used for either intolerance or lack of effectiveness within the 28 days after diagnosis of malaria.

Secondary outcome: parasitological cure rate at J3, fever clearance, digestive tolerance, number of relapses.

Design: Multicentric, open-label, randomized, controlled trial of superiority in adults with uncomplicated malaria and no contraindications to the oral treatment. Treatment will be administered for 3 days, and patients will be followed for 28 days, according to the national recommendations, to evaluate the therapeutic evolution. 640 patients will be included within 36 months. Recruitment will take place among 15 of the corresponding centres of the Malaria National Reference Centre.

Inclusion criteria : subjects aged more than 18, back from an endemic area with a positive diagnosis of Plasmodium falciparum by microscopic blood (thin and thick film) examination, able to come back at J3, J7 and J28, consent to participate.

Non inclusion criteria: pregnancy, ECG abnormality, contraindication to treatment, previous anti-malaric treatment within 30 days (HALOFANTRIN) or 48 hours (other antimalarial treatments).

Sample size justification: considering that 13% of patients on Malarone® will be treated by a second line of treatment, 300 patients per group would be necessary to achieve a relative reduction of 50% of patients treated by a second line of treatment (i.e. 6,5%) in the RIAMET® group, with a 80% of statistical power and a type I error rate taken to be 0,05. Considering 5% of patients lost of follow up, 640 patients have to be included.

Perspectives : these data should help to define the best 1st line of treatment in the uncomplicated malaria.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged more than 18,
* back from an endemic area with a positive diagnosis of Plasmodium falciparum by microscopic blood (thin and thick film) examination,
* absence of any severe manifestation according to the WHO definition of severe falciparum malaria

EXCLUSION CRITERIA:

* pregnancy,
* ECG abnormality,
* contraindication to treatment,
* previous anti-malaric treatment within 30 days,
* unable to come back at J3, J7 and J28,
* unwilling to consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2010-07; Primary Completion 2014-04 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of cases where a second line treatment is used for either intolerance or lack of effectiveness | within the 28 days after diagnosis of malaria

SECONDARY OUTCOMES:
Parasitological cure rate | At day 3
Fever clearance | At day 3
Digestive tolerance | At day 3
Number of relapses | At day 3

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Bouchaud, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Avicenne, Bobigny, Seine St Denis, France